CLINICAL TRIAL: NCT07394465
Title: First Tones: Artistic Communal Practices for 4 and 5 Year Old Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Collaborators: Federal University of Mato Grosso (Other); Universidade Federal do ABC (Unknown)
Responsible Party: Principal Investigator, Mayron Piccolo, Lecturer in Psychology, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB24-0032
Record Dates: First submitted 2026-01-23; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Mental Health
Keywords: Mental health; Preschoolers; Music based intervention; Singing; Communal music
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communal Singing (Experimental): Weekly music-based intervention including communal singing and rhythmic practices.
  Interventions: Behavioral: Communal singing
- Drawing (Active Comparator): Control condition involving drawing in a group while passively listening to the songs worked in the experimental condition.
  Interventions: Behavioral: Drawing

INTERVENTIONS:
Behavioral: Communal singing — The intervention group will participate in communal music sessions over a period of 10 weeks, once a week, after school. During this time, children will engage in age-specific communal music interventions, and sessions will be recorded on video.
  Other Names: Rhythmic exercises
  Arms: Communal Singing
Behavioral: Drawing — The control group will participate in drawing sessions over a period of 10 weeks, once a week. During this time, children will engage in artistic drawing activities while listening to the same music worked on in the intervention group, without, however, singing them together.
  Arms: Drawing

SUMMARY:
This project aims to develop therapeutic communal music interventions to support the mental health of preschool-aged children, identifying the psychological and neural mechanisms underlying these effects and comparing brain responses to communal versus non-communal music. The central hypothesis is that group musical practice will strengthen mental health indicators, promoting a sense of belonging and stimulating brain areas associated with reward. Communal singing interventions are economically viable and have demonstrated significant benefits in several populations. The research intends to fill gaps in the literature by identifying psychological mechanisms underlying the benefits of music and developing an assessment tool for the sense of belonging in preschoolers. Innovation also lies in exploring the emerging concept of communal music. The study will involve 30 children between the ages of 4 and 5, divided into an intervention group and a control group. Pre- and post-intervention assessments over a 10-week period will include behavioral, psychiatric, brain connectivity, and brain activity measures. In summary, this project seeks to develop accessible communal music interventions to enhance the mental health of 4- and 5-year-old children.

Our central hypothesis is that communal musical practice improves mental health markers in our sample by promoting a sense of belonging and differentially activating putative reward regions in the brain. By enhancing the sense of belonging and generating feelings of reward, we anticipate that the behavioral and psychiatric symptoms experienced by the target population will be attenuated. Our hypothesis was partially formulated based on recently obtained pilot data suggesting that communal music has protective effects against negative affect caused by ostracism, as well as literature on communal singing in other populations. The rationale for this proposed project is that understanding the therapeutic value of communal musical practice and identifying the mechanisms by which this occurs is likely to provide a strong scientific foundation for new strategies to support the mental health of at-risk groups and potentially reduce health disparities within these populations.

DETAILED DESCRIPTION:
This project aims to investigate the effects of a communal musical practice intervention on behaviors and neural markers of mental health in 4- and 5-year-old children. Children primarily search for emotional security, relational stability, and a sense of belonging from their immediate families, apart from school environments. Thus, there is great concern for children who experience family adversity and struggle to find belonging and stability at home.

A growing body of literature suggests that children who are born into dysfunctional, unstable family environments are at a much higher risk of future family instability, poorer life outcomes, and mental illness compared to children in more protected environments. Childhood adversity such as abuse, being raised in poverty, impaired parenting, etc., has been shown to drastically increase the likelihood of childhood mental disorders, behavioral problems, and subsequent depression in adulthood.

A relationship between lower socioeconomic position and experiencing childhood adversity has been found, and despite being at higher risk for the development of mental disorders, individuals in lower socioeconomic positions have reduced access to mental health treatment. Therefore, developing low-cost group-based interventions for children experiencing childhood adversity is of fundamental importance.

Communal singing interventions are low-cost and have shown significant benefits in other populations. For instance, Sung et al. explored the effects of a communal music intervention on anxiety and agitation symptoms in institutionalized older individuals with dementia. Individuals who participated in the 12-session intervention experienced a significant decrease in anxiety compared to those in a control group. Similarly, Adery and Park reported lower depression scores in individuals with psychiatric symptoms, namely psychosis and depression, who underwent a one-hour, eight-week communal singing intervention. Although no difference was seen for psychotic symptoms, individuals reported lower levels of loneliness, which could help explain some of the mechanisms through which communal music-making improves mental health.

Neuroimaging studies have shown significant changes in brain activity and connectivity following music-based interventions. For example, Quinci et al. reported increased functional connectivity between a mask containing auditory processing regions (e.g., superior temporal gyrus, middle temporal gyrus, and Heschl's gyrus) and the medial prefrontal cortex (mPFC) following intervention. These results are promising because the mPFC, for example, has been shown to be implicated in the maintenance of psychiatric disorders such as depression and post-traumatic stress disorder (PTSD). Furthermore, the mPFC is associated with reward processing. Interestingly, investigating reward-related processes has helped explain the pathophysiology of many psychiatric disorders.

Improving reward processing may be one of the mechanisms through which communal music-making improves mental health. Music listening has been associated with reward responses in the brain, and exploring the interaction between communal music-making, reward processing, and mental health markers warrants investigation. For instance, current promising interventions for some psychiatric disorders focus on improving reward processing as a means to decrease symptoms.

Building a sense of belonging may also be a mechanism involved in communal music-making. Besides the decreased loneliness experienced by individuals with psychosis following a choir-singing intervention, suggesting that singing together increased their sense of being connected to others, one qualitative study with individuals suffering from PTSD who underwent a communal music-making intervention that included communal performances reported an increased sense of belonging as well as self-confidence following intervention. Furthermore, in another qualitative study investigating the effects of communal singing in individuals with different mental disorders, Dingle et al. report increased feelings of connectedness to other members of the choir and the community in general. Finally, singing together also increases the levels of oxytocin, an important mediator of social behavior. Like reward processing, understanding the role of the sense of belonging in communal music-making warrants investigation.

ELIGIBILITY:
Inclusion Criteria:

* Age Group: Children who are 4 and 5 years old throughout the duration of the study will be included in the research.
* Interest: The child expresses a desire to participate in artistic activities.
* Informed Consent: Parents or legal guardians of children must provide informed consent for the children's participation in the project.
* Availability to participate: Children must be available and willing to participate in all activities.

Exclusion Criteria:

* Age outside the age range: Children outside the age range of 48 and 60 months will be excluded from the study.
* Lack of Consent: If parents or guardians do not agree to provide informed consent for the children's participation, they will be excluded from the study.
* Pre-existing Health Conditions: Children with health conditions that could significantly interfere with participation in activities, such as serious neurological disorders, serious mental disorders, or medical problems that contraindicate participation, will be excluded. This data will be collected in the registration form through a declaration from the child's parent or guardian. As a way of guaranteeing the anonymity of the research participant, all data collected will be carried out using an ID that will be linked to the participant's name. The name and respective ID will only be recorded on paper, which will be stored in a locked cabinet with access restricted to the responsible researcher.
* Participation in Simultaneous Activities: Children who are participating in other music teaching activities simultaneously that may interfere with the objectives or activities of this project will be excluded.
* Inability to Tolerate Activities: If a child demonstrates this during the familiarization session or at any time during the study, a significant inability to tolerate the proposed activities, including music lessons, playful quizzes, or the use of functional near-infrared spectroscopy (fNIRS), will be excluded.
* Non-Availability: If a child is not available to participate in all sessions or they and their guardians refuse to participate in any phase of the study, they will be excluded. The child is expected to attend all sessions.
* Incomplete Information: If parents or guardians do not provide complete and accurate information in the initial questionnaires, the child will be excluded from the study.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Child Behavioral Checklist 1.5-5 Total Score | Pre-test measures taken up to one day before the beginning of the intervention. Post-test measures taken starting the day to follow the last session until one month following completion (10 weeks)
  Developed by Achenbach and Rescorla, with studies in the Brazilian context indicating good reliability, this instrument seeks to obtain standardized measures of emotional and behavioral problems in preschool children, based on parent reports. It consists of 99 items, responded to on a 3-point likert scale (0 = not true, 1 = somewhat or sometimes true, 2 = very true or often true).

SECONDARY OUTCOMES:
Internalized Symptoms | Pre-test measures taken up to one day before the beginning of the intervention. Post-test measures taken starting the day to follow the last session until one month following completion (10 weeks)
  This scale will come from the Child Behavior Checklist 1.5-5 and will include the following sub scales: emotional reactivity, anxiety/depression, somatic complaints, withdrawn behavior.
Externalizing Symptoms | Pre-test measures taken up to one day before the beginning of the intervention. Post-test measures taken starting the day to follow the last session until one month following completion (10 weeks)
  These will come from the following sub scales of the Child Behavior Checklist 1.5-5: attention problems, and aggressive behavior.

OTHER OUTCOMES:
Subscales of the Child Behavior Checklist 1.5-5 | Pre-test measures taken up to one day before the beginning of the intervention. Post-test measures taken starting the day to follow the last session until one month following completion (10 weeks)
  Emotional reactivity, anxiety/depression, somatic complaints, withdrawn behavior, attention problems, aggressive behavior, and sleep problems.

CONTACTS AND LOCATIONS:
Overall Officials: Mayron Piccolo, PhD, Principal Investigator — Harvard University
Locations (2):
- Brazil (2):
  - Universidade Federal de Mato Grosso do Sul, Campo Grande, Mato Grosso do Sul
  - Universidade Federal do ABC Paulista, São Bernardo do Campo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lam CF, Caterina P, Filion P, van Heerden PV, Ilett KF. The ratio of polymorphonuclear leucocytes (PMN) to non-PMN cells--a novel method of assessing acute lung inflammation. Exp Toxicol Pathol. 2002 Nov;54(3):187-91. doi: 10.1078/0940-2993-00250. PMID 12484554
- See also: Study Page — https://mpiccolo.scholars.harvard.edu/communal-music-making-children-experiencing-familial-adversities